CLINICAL TRIAL: NCT01491880
Title: Feasible Delivery of CBT for Rural Latino Youth With Anxiety
Brief Title: Treatment Study for Rural Latino Youth With Anxiety
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH090149; R34MH090149 (NIH)
Record Dates: First submitted 2011-07-29; First posted 2011-12-14 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Anxiety Disorders; Separation Anxiety Disorder; Social Anxiety Disorder; Specific Phobia; Generalized Anxiety Disorder
Keywords: cognitive behavior therapy; telemedicine; rural; Latinos; children
MeSH Terms: conditions — Anxiety Disorders; Anxiety, Separation; Phobia, Social; Phobia, Specific; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child Anxiety Program by Telephone (Experimental): The child anxiety program by telephone is an adaptation of Ron Rapee's Cool Kids Outreach Program (Lyneham and Rapee, 2006) for child anxiety, with appropriate adaptations made to meet the needs of rural Latino families (including a Spanish translation). This is a parent mediated program, where parents are taught how all the skills of cognitive behavior therapy (CBT) and how to apply these skills to these children's anxieties. Children are also expected to participate, however all direct contact that a therapist may have, is with the parent only.
  Interventions: Behavioral: Therapist-Assisted by Telephone
- Child Anxiety Program- Self Help (Experimental): Families randomized to the Self-Help CBT condition will receive program materials along with instructions for completing weekly assignments. Specifically, they will receive the same materials as families in the telephone-based condition however in the self-help group, parents and children are expected to read the materials for that week and complete the workbook activities without planned therapist involvement. Instead they will be given the option to initiate a telephone call to the therapist, if they have questions or need extra support.
  Interventions: Behavioral: Self-Help

INTERVENTIONS:
Behavioral: Therapist-Assisted by Telephone — Parents will receive educational workbooks and ongoing support over the phone from a child anxiety specialist to learn how to use cognitive behavioral therapy skills to manage their children's fears and worries.
  Arms: Child Anxiety Program by Telephone
Behavioral: Self-Help — Parents will receive educational workbooks to learn how to use cognitive behavioral therapy skills to manage their children's fears and worries independently. Parents will have the option to access support over the phone from a child anxiety specialist.
  Arms: Child Anxiety Program- Self Help

SUMMARY:
This pilot study will examine the feasibility of two modes of service delivery (e.g., a minimal therapist contact, self-help program, and a more intensive therapist supported, telephone-based approach) in a rural, primarily Latino, population. These modes of delivery may ultimately improve access to evidence based treatments and mental health outcomes among underserved groups.

DETAILED DESCRIPTION:
Children with anxiety disorders are often characterized by an unmet need for treatment however, in special populations such as Latino and rural youth, such disparities are compounded by the effects of culture and geographic isolation. More specifically, barriers related to language, stigma, and access often lead to lower rates of utilization and poorer outcomes among children in need of mental health services (Alvidrez and Azocar, 1999; McCabe et al., 2002; Myers et al., 2008; Vega et al., 2001). These findings are disappointing given abundant data supporting the effectiveness of cognitive behavior and behavior therapies for children with anxiety disorders (Barrett et al., 1996; Beidel et al., 2007; Kendall & Southam-Gerow, 1996; Walkup et al., 2008). Efforts to examine feasible methods to deliver evidence-based treatments to children with anxiety disorders are critical in order to extend quality care to underserved groups. The goal of this R34 is to address these disparities, by translating and tailoring an existing child anxiety cognitive behavior therapy program (The Cool Kids Outreach Program; Lyneham and Rapee, 2006), to fit the needs of Spanish-speaking rural families and examining the feasibility, acceptability, tolerability and safety of implementing this intervention using varying modes of delivery.

A pilot study for children (age 8-13) with anxiety disorders (i.e., separation anxiety disorder, generalized anxiety disorder, social anxiety disorder, and specific phobias) will be conducted and 40 children will be randomized to two service delivery modes which represent varying levels of therapist contact: 1) 20 families will be randomized to a telephone-based, therapist-supported CBT program, and; 2) 20 families will be randomized to a more minimal contact bibliotherapy condition (primarily CBT self-help materials). All families will be recruited from primary care settings, given its defacto mental health service status. Feasibility and clinical outcomes will be measured at baseline, midtreatment and post-treatment. Additionally, during exit interviews, participants (as well as those who may have dropped out of the program) will be asked to discuss the perceived usefulness, acceptability, and impact of the intervention. This pilot study will provide important data regarding the feasibility, acceptability, tolerability and safety of the intervention conditions as well as the opportunity to pilot procedures that will be used in a larger effectiveness trial with rural Latino youth.

ELIGIBILITY:
Inclusion Criteria:

* Child between ages of 8-13
* Meets DSM-IV criteria for one of the following disorders: separation anxiety disorder, social phobia, generalized anxiety disorder, specific phobia, or obsessive-compulsive disorder
* If takes a medication, has maintained a stable dose for 3 months before baseline assessment
* Pediatric medical care is provided through one of the participating primary care clinics
* Parent and child are fluent in English or Spanish
* Family has easy access to a telephone

Exclusion Criteria:

* Comorbid diagnosis, such as major depression, ADHD, or psychosis that is considered clinically significant and the primary problem
* Life threatening conditions, active suicidality, psychotic disorders, bipolar disorder or pervasive developmental disorders

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Consumer Satisfaction Questionnaire | Pre-treatment and Post-treatment (maximum of 6 months after randomization)
  The aim of this pilot study is to understand issues of feasibility rather than formal hypothesis testing.
  The construct of acceptability will be evaluated by parents' reports on Consumer Satisfaction Questionnaire (March et al., 1999). Overall mean scores reflecting at least "above average" ratings (5 or greater on Consumer Satisfaction) will be considered acceptable.

SECONDARY OUTCOMES:
Barriers to Treatment Participation Scale | Pretreatment & Posttreatment (maximum of 6 months after randomization)
  Overall feasibility will be defined as the ability to complete the study procedures and goals in the proposed time frame. Further the feasibility of the program will be evaluated by participants' report on the Barriers to Treatment Participation Scale (Kazdin et al., 1997); overall mean scores reflecting that "barriers" were "never a problem, occasionally a problem or sometimes a problem" will be considered acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Chavira, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Chavira DA, Bustos C, Garcia M, Reinosa Segovia F, Baig A, Ng B, Camacho A. Telephone-assisted, parent-mediated CBT for rural Latino youth with anxiety: A feasibility trial. Cultur Divers Ethnic Minor Psychol. 2018 Jul;24(3):429-441. doi: 10.1037/cdp0000186. Epub 2018 May 24. PMID 29792485